

# LONG-TERM SEQUELAE OF COVID-19 (MYALGIC ENCEPHALOMYELITIS: AN INTERNATIONAL CROSS-SECTIONAL STUDY

GLOBAL LONG COVID STUDY BY ICRAAA TEAM

| Contents |
|---|
| Collaborating with International Clinical Research Association & Allied Activities (ICRAAA) |
| ACTIVITIES OF THE ASSOCIATION |
| Protocol summary |
| Study Title |
| Introduction |
| Aim |
| Objectives |
| Study Design4 |
| Study duration4 |
| What are the study procedures? |
| What type of questions will be asked?5 |
| Who can fill the survey? (inclusion/exclusion criteria)5 |
| Are there any risks to participating in this study?5 |
| What are the benefits for participating in this study?5 |
| Can participants choose to leave the study?6 |
| How will participants' information be kept confidential? |
| Are participants paid to be in this study?8 |
| Whom do participants contact for questions? |
| Financial support: |
| Authorship & collaboration |

| erences: |
|----------|
|----------|

Collaborating with International Clinical Research Association & Allied Activities (ICRAAA) International Clinical Research Association & Allied Activities (ICRAAA) is an international group based in Alexandria, Egypt meant by clinical, research primary and secondary. The association was founded on April 20, 2021, by Ahmed Shaheen, a 4th-year medical student at Alexandria faculty of medicine. The Association has its internal structure composed of a president, two vice presidents, three coordinators, and one honorable president.

The main goal of the association is to provide a real opportunity and suitable atmosphere for medical students, new graduates, and physicians from all over the world to start their career in clinical research. We have two parallel goals training the beginners and providing the right experts in the field you are interested in to help in your research project. We are more concerned about members from low- and middle-income countries because of the lack of real training in medical research and lack of funding which is a major problem for both medical students and new graduates who consider a future career in medical research.

#### **ACTIVITIES OF THE ASSOCIATION**

- 1. Conducting clinical research primary and secondary research. 2. Holding research training sessions and journal clubs.
- 3. An annual conference mainly for work produced by the association, it will be either virtual or in-person at Alexandria

city, Egypt. 4. Targeting to have our scientific journal. (long-term objective) 5. Gathering emerging researchers from lowand middle-income countries together in one place to guarantee better interaction, cooperation, and learning from different experiences.

6. We will open a call for a Research training scholarship every 6 months.

## Protocol summary

| Study Title | Long-term sequelae COVID-19 (Myalgic encephalomyelitis: an international cross-sectional study |
|---|---|
| | Novel COVID-19 pandemic caused by SARS-CoV-2 have a lot |
| Introduction | of serious symptoms, but some of last for a period of time even |
| | after the recovery. Even people who had some mild symptoms |
| | during COVID-19 continue to have long terms effects after |
| | initial recovery. These people are called "long haulers" and |
| | these symptoms are called Long COVID-19, so in this study, we |
| | aim to detect the most common symptoms of long Covid_19 |
| | syndrome |

| Aim | This study aims to provide a comprehensive global picture of the post covid symptoms and the potential Myalgic encephalitis cases incidence |
|---|---|
| Objectives | The primary objective of this research is to understand acute |
| | and chronic long covid symptoms by asking questions detecting |
| | patient's experience especially symptoms lasting for several |
| | months which is known as chronic fatigue syndrome(Myalgic |
| | encephalitis). The study focuses on symptoms describing |
| | Myalgic encephalitis which may still affect covid patients for |
| | several months after the infection along with making a big |
| | picture about rare symptoms that may the patient experienced |
| | during or after the infection. |
| | A secondary objective of this research is to focus on the long- |
| | term sequelae effects and comorbidities following COVID-19 |
| | vaccination. |
| Study Design | cross sectional online-questionnaire based study. |
| Study duration | |

| What are the study procedures? | If you agree to participate after reading this message, you will |
|---|---|
| | be taken to the survey which is housed on the Survey Heart |
| | platform. You will be asked to answer the questions to the best |
| | of your ability. In the mental health section and any question |
| | marked as optional, you can choose whether or not you would |
| | like to respond. The information that you enter will be collected |
| | after each page. You can take breaks and return to finish the |
| | survey at any time within one week. |
| What type of questions will be asked? | The survey asks different questions on testing, diagnosis, |
| | symptoms, treatments, background information, coping |
| | methods as well as health and mental health. |
| | Persons had a COVID-19, or suspected COVID-19 |
| Who can fill the survey? (inclusion/exclusion criteria) | infection (still suffering or suffered symptoms) for longer |
| | than 1 week Even if your COVID-19 test result was |
| | negative, or you were not tested at all |
| | Persons who are 18 years of age or older |
| Are there any risks to participating in this study? | There are no known risks associated with this research study. In |
| , | order to mitigate risks inherent in all online surveys, this survey |
| | will be conducted on the Survey Heart platform. |
| What are the benefits for participating in this study? | There are no known direct benefits associated with participating |
| | in this research study. Your experiences will help us to better |
| | define the recovery from the COVID19 and improve advocacy |
| | for Long COVID (long-hauler) population |

| Can participants choose to leave the study? | Participation in this study is voluntary. You may refuse to participate or at any point during the survey, if you decide to opt out from our study, you can fill this form by providing the anonymous ID we generate for you. Once you submit the survey you will be unable to withdraw your data. |
|---|---|

How will participants' information be kept confidential?

There will be no information collected that may in any way identify you based upon your responses Email addresses will only be used to send you a link to the survey, or to notify you of future surveys. A cryptographic algorithm will be used to generate a hash code from each email address. Hash codes will link survey responses to a unique participant without revealing the participant's email address or identity. Paired email addresses and hash codes will be stored in a GDPR compliant email database managed by a secure hosting provider. Survey responses will be stored on a separate server in a secure, encrypted format. Email addresses will not be stored with survey responses and will remain unknown to both the research team and the hosting company. Any data exported will only be used by the above survey investigators and exported data will be housed solely on secure servers.

Your responses will be housed on a secure server for 10 years, after which they will be destroyed. Anonymized data may be made public or shared with any other researchers.

| Are participants paid to be in this study? | You will receive no monetary compensation or gifts for participating in this study. |
|---|---|
| Whom do participants contact for questions? | If you have any questions about the study, please contact ICRAAACovid@gmail.com Please note that email is not a secure form of communication. |
| Financial support: | self-funding |
| Authorship& collaboration | |

### References:

1. WHO Coronavirus (COVID-19) Dashboard | WHO Coronavirus (COVID-19) Dashboard With Vaccination Data [Internet]. [cited 2021 Sep 10]. Available from: https://covid19.who.int/

- 2. Komaroff AL, Bateman L. Will COVID-19 Lead to Myalgic Encephalomyelitis/Chronic Fatigue Syndrome? Frontiers in Medicine. 2021 Jan 18;0:1132.
- 3. Crook H, Raza S, Nowell J, Young M, Edison P. Long covid—mechanisms, risk factors, and management. BMJ. 2021 Jul;374:n1648.
- 4. Carfì A, Bernabei R, Landi F. Persistent symptoms in patients after acute COVID-19. JAMA Journal of the American Medical Association. 2020 Aug;324(6):603–5.
- 5. MW T, SS K, CJ L, E BR, NI S, DC F, et al. Symptom Duration and Risk Factors for Delayed Return to Usual Health Among Outpatients with COVID-19 in a Multistate Health Care Systems Network United States, March-June 2020. MMWR Morbidity and mortality weekly report. 2020 Jul;69(30):993–8.
- 6. Carruthers BM, Sande MI van de, Meirleir KL de, Klimas NG, Broderick G, Mitchell T, et al. Myalgic encephalomyelitis: International Consensus Criteria. Journal of Internal Medicine [Internet]. 2011 Oct 1 [cited 2021 Sep 10];270(4):327–38. Available from: https://onlinelibrary.wiley.com/doi/full/10.1111/j.1365-2796.2011.02428.x
- 7. Coronavirus disease (COVID-19): Vaccines safety.
- 8. Alobaida S, Lam JM. Beau lines associated with COVID-19. CMAJ [Internet]. 2020 Sep 8 [cited 2021 Sep 10];192(36):E1040–E1040. Available from: https://www.cmaj.ca/content/192/36/E1040
- 9. Sperber AD. Translation and validation of study instruments for cross-cultural research. Gastroenterology [Internet]. 2004 Jan 1 [cited 2021 Sep 10];126(1):S124–8. Available from: http://www.gastrojournal.org/article/S0016508503015646/fulltext

Thank you for joining the Global Long covid study by ICRAAA. For any questions or suggestions, don't hesitate to contact us at:

Email: ICRAAACovid@gmail.com